CLINICAL TRIAL: NCT01941680
Title: Observational Prospective Study, Evaluating the Standard of Care as Recommend by International Consensus With Zidovudine-Pegylated Interferon +/-Polychemotherapy in High Risk Adult-T-cell Lymphoma/Leukaemia (T-cell Lymphoma/Leukaemia) Followed by Allogeneic Transplant Among Eligible Patients Younger Than 65 Years Old
Brief Title: High Risk Adult T-cell Leukemia/Lymphoma (ATLL-HR) and Allogeneic Transplant
Acronym: ATLL-HR-01
Status: Completed | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 13/B/04; 2013-A00327-38 (Other: AFSSAPS)
Record Dates: First submitted 2013-09-03; First posted 2013-09-13 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: T-cell Lymphoma; Leukaemia
MeSH Terms: conditions — Lymphoma, T-Cell; Leukemia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- ZPI: Zidovudine 1000mg/day : Retrovir® 250mg/day) PegINF (Pegasys®) 180μg x1 injection/week
- ZPI+CHOP-21: Zidovudine 1000mg/day : Retrovir® 250mg/day) PegINF (Pegasys®) 180μg x1 injection/week
  CHOP-21 Day1 = day 21 (3 cycles)
  Day 1 Cyclophosphamide : 750 mg/m2, Doxorubicine : 50 mg/m2, Vincristine : 1,4mg/m2, Prednisone : 100mg/day PO.
  day 2-Day 5 Prednisone
  1mg/kg/day PO.
- ZPI +DHAP-21: Zidovudine 1000mg/day : Retrovir® 250mg/day) PegINF (Pegasys®) 180μg x1 injection/week
  DHAP Day 1= day 21 (3 cycles) Day 1 : Cisplatina 100 mg/m2 Day 2 and day 3 : Aracytine 2000mg/m2/day Day 1-day 4 : Dexamethasone 40mg

SUMMARY:
Patients are recruited at diagnosis or at relapse of ATLL-HR in French Caribbean islands and Guyana. They all receive Zidovudine and Pegylated Interferon (ZPI). For patients younger than 65 years old, an allogeneic donor is searching out. Patients included at relapse and with lymphoma clinico-biological subtype also receive chemotherapy (CT). Responses are assessed during ZPI+/-CT and eligible patients (depending on age, comorbidities and response criteria) receive allogeneic transplant. Patient follow-up is planned for 3 years old

ELIGIBILITY:
Inclusion Criteria:

* Patient >18 years old and ≤ 75 years old, with ATLL-HR who signed informed consent.

Exclusion Criteria:

* Pregnant or nursing women are not eligible; neither are women of childbearing potential unless using effective contraception as determined by the patient's physician.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Populations of French Caribbean Islands and Guyana with ATLL-HR. .
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-10-31 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with relapse | Up to 3 year

SECONDARY OUTCOMES:
Evidence of presence of gene expression of Tax and HBZ confirmed by Rt-PCR | 1 year
  The titrations of genes are performed at month 12, month 24 and month 36

CONTACTS AND LOCATIONS:
Locations (2):
- CHU Pinteà Pitre/Abymes, Pointe-à-Pitre, Guadeloupe
- CHU de Martinique, Fort-de-France, Martinique